CLINICAL TRIAL: NCT00686309
Title: Comparison of On-line and Off-line Measurements of Exhaled NO
Brief Title: Comparison of On-line and Off-line Measurements of Exhaled Nitric Oxide (NO)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Israel Amirav, Ziv Medical center
Other Study IDs: HP8-295-R
Record Dates: First submitted 2008-05-26; First posted 2008-05-29 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Asthma; Primary Ciliary Dyskinesia
Keywords: exhaled NO; off line; on line; comparison; Bland altman method
MeSH Terms: conditions — Asthma; Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Asthma is a major health problem worldwide. The measurement of fractional exhaled nitric oxide (FENO) has been established as a valuable non invasive and simple tool in the diagnosis of asthma and may also act as a useful surrogate inflammatory marker on which to base treatment decisions in asthma management algorithms. The measurement is useful also in other respiratory diseases. Current methods of measuring FENO include on line measurements by heavy duty expensive analyzers which are not widely and easily available. Off line measurements of breath samples which can be analysed later may be a simple solution. We hypothesize tha toff line measurements of NO will be as reliable and valid as those measured on-line

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate
* Filed a short health questionnaire

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: General population bth healthy and with respiratory illness such as asthma, COPD, PCD, Rhinitis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Off line measurement of exhaled NO | Two types of breathing in the same day

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Department, Ziv Medical Center, Safed, Israel